CLINICAL TRIAL: NCT05967052
Title: Investigation of Pregabalin Therapy and Complex Rehabilitation in Treating Chronic Fatigue Associated With Post-COVID Syndrome
Brief Title: Investigation of Treating Chronic Fatigue Syndrome After COVID With Pharmacotherapy (Pregabalin) or Complex Rehabilitation
Acronym: POSTCOVID
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Geriatrics, Rheumatology and Rehabilitation, Poland (Network)
Collaborators: Medical Research Agency, Poland (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NIGRIR_001POSTCOVID
Record Dates: First submitted 2023-07-28; First posted 2023-08-01 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Chronic Fatigue Syndrome; COVID-19, Long Haul
Keywords: chronic fatigue syndrome; associated with post-COVID syndrome
MeSH Terms: conditions — Fatigue Syndrome, Chronic; Post-Acute COVID-19 Syndrome | interventions — Pregabalin; Telerehabilitation; Psychotherapy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Pregabalin (Experimental)
  Interventions: Drug: Pregabalin; Behavioral: Independent walking training
- Pregabalin + Rehabilitation (Experimental)
  Interventions: Drug: Pregabalin; Behavioral: Independent walking training; Behavioral: Gradual movement therapy in the ward; Behavioral: Telerehabilitation; Behavioral: Psychotherapy
- Rehabilitation + Placebo (Experimental)
  Interventions: Behavioral: Independent walking training; Drug: Placebo; Behavioral: Gradual movement therapy in the ward; Behavioral: Telerehabilitation; Behavioral: Psychotherapy
- Placebo (Placebo Comparator)
  Interventions: Behavioral: Independent walking training; Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Pregabalin pharmacotherapy
  Arms: Pregabalin; Pregabalin + Rehabilitation
Behavioral: Independent walking training — Independent walking training
Drug: Placebo — Placebo
  Arms: Placebo; Rehabilitation + Placebo
Behavioral: Gradual movement therapy in the ward — Gradual movement therapy in the ward
  Arms: Pregabalin + Rehabilitation; Rehabilitation + Placebo
Behavioral: Telerehabilitation — Telerehabilitation
  Arms: Pregabalin + Rehabilitation; Rehabilitation + Placebo
Behavioral: Psychotherapy — Psychotherapy
  Arms: Pregabalin + Rehabilitation; Rehabilitation + Placebo

SUMMARY:
This is a single-center, prospective, randomized, double-blind (pharmacotherapy), placebo-controlled, and comprehensive rehabilitation phase II clinical trial to determine the usefulness of pregabalin in a new indication (post-COVID chronic fatigue syndrome).

Patients will be randomized in a 1:1:1:1 ratio to pregabalin (75-300 mg daily in two divided doses), comprehensive rehabilitation with a placebo drug, comprehensive rehabilitation with pregabalin (75-300 mg in two divided doses), or placebo (two divided doses) for 6 months (177-187 days).

There will be 4 outpatient visits to the research center and 12 telephone consultations.

The procedures and assessments performed as part of the study are listed in the study schedule.

It is planned to include 132 patients in the study, which, assuming a 10% level of non-completion of the program, will result in the examination of 120 patients (30 in each arm).

Patients will be recruited during an outpatient medical consultation with a general practitioner or neurologist, psychiatrist, psychologist or other specialists, as well as with the use of information materials in the form of leaflets and advertisements on the Internet.

ELIGIBILITY:
Inclusion Criteria:

1. The patient correctly gave written informed consent to participate in the study;
2. Men or women between the ages of 18 and 65 inclusive at the time of signing the informed consent;
3. Patient after a minimum of 6 months from the documented detection of SARS-CoV-2 infection (document confirming the history of the disease, including a positive result of the PCR or antigen test, certificate of convalescence; medical documentation confirming the infection; the condition is also considered fulfilled in the case of documented infection asymptomatic);
4. During the screening, the patient meets the criteria for the diagnosis of chronic fatigue syndrome (CFS) according to the National Academy of Medicine (2015);
5. Women:

   a) incapable of having children (post-menopausal or child-bearing, subjected to permanent sterilization); (b) of childbearing potential with a negative pregnancy test result at screening and using a highly effective method of contraception throughout the IMP use and for 7 days after the last IMP use.
6. The patient agrees to participate in all activities provided for in the study.
7. The patient is able to understand the information presented and give informed consent to participate in the study prior to screening.

Exclusion Criteria:

1. Vital functions disorders;
2. Documented hypersensitivity to pregabalin or any of the excipients of the formulation (i.e., lactose);
3. Moderate or severe depression during treatment or present during psychiatric evaluation at baseline;
4. Concurrent treatment with opioids or other antiepileptic drugs (including tramadol, buprenorphine, morphine, oxycodone, gabapentin, duloxetine);
5. Pregnant or breastfeeding women.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Change in fatigue intensity expressed as a difference in Multidimensional Fatigue Inventory-20 (MFI-20) score | 3 months and 6 months
  Change in fatigue intensity expressed as a difference in Multidimensional Fatigue Inventory-20 (MFI-20) score at 3 and 6 months of the study relative to the baseline score
Walking distance as a difference in score from the 6 Minute Walking Test | 3 months and 6 months
  Walking distance as a difference in score from the 6 Minute Walking Test at 3 and 6 months compared to baseline

SECONDARY OUTCOMES:
Change in the level of satisfaction with life expressed in the form of the result of the Satisfaction with Life Scale (Juczyński) | 3 months and 6 months
  Change in the level of satisfaction with life expressed in the form of the result of the Satisfaction with Life Scale (Juczyński) in the 3rd and 6th month of the study in relation to the result on the day of the study
Change in the result obtained in the "Beck Depression Inventory (BDIII)" study | 3 months and 6 months
  Change in the result obtained in the "Beck Depression Inventory (BDIII)" study in the 3rd and 6th month of the study in relation to the result on the day of the study commencement.
Change in the result obtained in the anxiety test - State and Trait Anxiety Inventory (STAI) | 3 months and 6 months
  Change in the result obtained in the anxiety test - State and Trait Anxiety Inventory (STAI) in the 3rd and 6th month of the study in relation to the result on the day of the study commencement.
Change in the degree of acceptance of the disease assessed by the Acceptance of Illness Scale (Juczyński) i | 3 months and 6 months
  Change in the degree of acceptance of the disease assessed by the Acceptance of Illness Scale (Juczyński) in the 3rd and 6th month of the study in relation to the result on the day of starting the study
Change in the result of the CCT test | 3 months and 6 months
  Change in the result of the CCT test in the 3rd and 6th month of the study compared to the result on the day of starting the study.
Change in neuropsychological assessment expressed by the change in the result of the Wisconsin Card Sorting Test (WCST) | 3 months and 6 months
  Change in neuropsychological assessment expressed by the change in the result of the Wisconsin Card Sorting Test (WCST) in the 3rd and 6th month of the study compared to the result on the day of the study commencement.
Change in the result of the RFFT test | 3 months and 6 months
  Change in the result of the RFFT test in the 3rd and 6th month of the study compared to the result on the day of starting the study.
Change in the WAIS-R intelligence test result | 3 months and 6 months
  Change in the WAIS-R intelligence test result in the 3rd and 6th month of the study in relation to the result on the day of the study commencement
Change in reaction time expressed by the Stroop interference test | 3 months and 6 months
  Change in reaction time expressed by the Stroop interference test in the 3rd and 6th month of the study compared to the result on the day of the study start.
Change in the assessment of the quality of gait | 3 months and 6 months
  Change in the assessment of the quality of gait in the 3rd and 6th month of the study in relation to the result on the day of the beginning of the study
Change in walking speed | 3 months and 6 months
  Change in walking speed in the 3rd and 6th month of the study in relation to the result on the day of the study.

OTHER OUTCOMES:
The change in the profile of the examined inflammatory cytokines | 3 months and 6 months
  The exploratory endpoint is the change in the profile of the examined inflammatory cytokines in the 3rd and 6th month of the study in relation to the result before the start of the study.
Number of adverse events and the number and percentage of patients who experienced adverse events | 3 months and 6 months
  Number of adverse events and the number and percentage of patient who experienced adverse events
Number of adverse events and the number and proportion of patients who experienced treatment-related adverse events | 3 months and 6 months
  Number of adverse events and the number and proportion of patients who experienced treatment-related adverse events
Number of serious adverse events and number and proportion of patients with serious adverse events. | 3 months and 6 months
  Number of serious adverse events and number and proportion of patients with serious adverse events.
Number of serious adverse events and the number and proportion of patients who experienced treatment-related serious adverse events. | 3 months and 6 months
  Number of serious adverse events and the number and proportion of patients who experienced treatment-related serious adverse events.
Number and percentage of patients who discontinued participation in the study due to an adverse event - changes in laboratory parameters and basic vital signs. | 3 months and 6 months
  Number and percentage of patients who discontinued participation in the study due to an adverse event - changes in laboratory parameters and basic vital signs.

CONTACTS AND LOCATIONS:
Overall Officials: Beata Tarnacka, Prof, Md, PhD, Principal Investigator — National Institute of Geriatrics, Rheumatology and Rehabilitation
Locations (1):
- Centrum Wsparcia Badań Klinicznych, Warsaw, Masovian Voivodeship, Poland